CLINICAL TRIAL: NCT01180452
Title: Endoscopic Detection of Small Bowel Dysplasia and Cancer in Patients With Jejuna or Ileal Crohn Disease : Prospective Study in a Cohort of High Risk Patients
Brief Title: Endoscopic Detection of Dysplasia in Crohn 's Disease Patient
Acronym: DYDJI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GETAID 2008-4
Record Dates: First submitted 2010-03-31; First posted 2010-08-12 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Crohn Disease Located in Jejunum or Ileum
Keywords: Crohn disease; dysplasia; adenocarcinoma; endoscopy; jejunum; ileum
MeSH Terms: conditions — Crohn Disease; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group open label (Other): Prospective Cohort
  Interventions: Procedure: enteroscopy

INTERVENTIONS:
Procedure: enteroscopy — endoscopic enteroscopy to do biopsies on jejunum

SUMMARY:
Patients with Crohn's disease (CD) have an increased risk of small bowel adenocarcinoma (SBA). Long duration of CD is the main risk factor. SB dysplasia has been associated with SBA in 20% of cases, always described in diseased sites. The progression to neoplasia and natural history remains unknown but progression of inflammation to dysplasia and then to adenocarcinoma is suspected.

As for surveillance recommendations for colorectal carcinoma in long standing inflammatory colonic disease, endoscopic screening of SB could be proposed in CD patients with risk factors of SBA. No study can be found in literature.

The investigators propose a multicenter exploratory open study on prospective cohort of CD patients with high risk of dysplasia or cancer. The goal is evaluate the rate of dysplasia and adenocarcinoma detected by enteroscopy with biopsies in a high risk CD population

ELIGIBILITY:
Inclusion Criteria:

* More than 18-years-old
* Crohn disease on jejunum and/or ileum since at least 10 years
* Radiography done during last year

Exclusion Criteria:

* Dysplasia previously detected
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Frequency of dysplasia and adenocarcinoma | 2 months
  dysplasia will be described as high or low level Samples will be analysed by 2 different team of anapathologists

SECONDARY OUTCOMES:
Success of endoscopic detection | 1-3 Months
  the success will be measured by reaching at least one pathologic area during the endoscopic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marion Simon, Doctor, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Marc Lémann, PhD, Study Chair — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Yoram BOUHNIK, PhD, Study Director — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (15):
- France (15):
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - Hopital Beaujon, Clichy
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - Chru Lille, Lille
  - CHU NICE, Nice
  - Hopital Saint Louis, Paris
  - Institut Mutualiste Montsouris (Imm), Paris
  - Hopital Haut Leveque, Pessac
  - CHU LYON, Pierre-Bénite
  - Chu Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours
  - Chu Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Abrahams NA, Halverson A, Fazio VW, Rybicki LA, Goldblum JR. Adenocarcinoma of the small bowel: a study of 37 cases with emphasis on histologic prognostic factors. Dis Colon Rectum. 2002 Nov;45(11):1496-502. doi: 10.1097/01.DCR.0000034134.49346.5E. PMID 12432298
- [Result] von Roon AC, Reese G, Teare J, Constantinides V, Darzi AW, Tekkis PP. The risk of cancer in patients with Crohn's disease. Dis Colon Rectum. 2007 Jun;50(6):839-55. doi: 10.1007/s10350-006-0848-z. PMID 17308939
- [Result] Jess T, Gamborg M, Matzen P, Munkholm P, Sorensen TI. Increased risk of intestinal cancer in Crohn's disease: a meta-analysis of population-based cohort studies. Am J Gastroenterol. 2005 Dec;100(12):2724-9. doi: 10.1111/j.1572-0241.2005.00287.x. PMID 16393226
- [Result] Canavan C, Abrams KR, Mayberry J. Meta-analysis: colorectal and small bowel cancer risk in patients with Crohn's disease. Aliment Pharmacol Ther. 2006 Apr 15;23(8):1097-104. doi: 10.1111/j.1365-2036.2006.02854.x. PMID 16611269
- [Result] Palascak-Juif V, Bouvier AM, Cosnes J, Flourie B, Bouche O, Cadiot G, Lemann M, Bonaz B, Denet C, Marteau P, Gambiez L, Beaugerie L, Faivre J, Carbonnel F. Small bowel adenocarcinoma in patients with Crohn's disease compared with small bowel adenocarcinoma de novo. Inflamm Bowel Dis. 2005 Sep;11(9):828-32. doi: 10.1097/01.mib.0000179211.03650.b6. PMID 16116317
- [Result] Lashner BA. Risk factors for small bowel cancer in Crohn's disease. Dig Dis Sci. 1992 Aug;37(8):1179-84. doi: 10.1007/BF01296557. PMID 1499440
- [Result] Solem CA, Harmsen WS, Zinsmeister AR, Loftus EV Jr. Small intestinal adenocarcinoma in Crohn's disease: a case-control study. Inflamm Bowel Dis. 2004 Jan;10(1):32-5. doi: 10.1097/00054725-200401000-00005. PMID 15058524
- [Result] Piton G, Cosnes J, Monnet E, Beaugerie L, Seksik P, Savoye G, Cadiot G, Flourie B, Capelle P, Marteau P, Lemann M, Colombel JF, Khouri E, Bonaz B, Carbonnel F. Risk factors associated with small bowel adenocarcinoma in Crohn's disease: a case-control study. Am J Gastroenterol. 2008 Jul;103(7):1730-6. doi: 10.1111/j.1572-0241.2008.01847.x. Epub 2008 Jun 28. PMID 18564124
- [Result] Yamamoto T, Fazio VW, Tekkis PP. Safety and efficacy of strictureplasty for Crohn's disease: a systematic review and meta-analysis. Dis Colon Rectum. 2007 Nov;50(11):1968-86. doi: 10.1007/s10350-007-0279-5. PMID 17762967
- [Result] Greenstein AJ, Sachar D, Pucillo A, Kreel I, Geller S, Janowitz HD, Aufses A Jr. Cancer in Crohn's disease after diversionary surgery. A report of seven carcinomas occurring in excluded bowel. Am J Surg. 1978 Jan;135(1):86-90. doi: 10.1016/0002-9610(78)90015-6. No abstract available. PMID 623378
- [Result] Ribeiro MB, Greenstein AJ, Heimann TM, Yamazaki Y, Aufses AH Jr. Adenocarcinoma of the small intestine in Crohn's disease. Surg Gynecol Obstet. 1991 Nov;173(5):343-9. PMID 1948581
- [Result] Watermeyer G, Locketz M, Govender D, Mall A. Crohn's disease-associated small bowel adenocarcinoma with pre-existing low-grade dysplasia: a case report. Am J Gastroenterol. 2007 Jul;102(7):1545-6. doi: 10.1111/j.1572-0241.2007.01166.x. No abstract available. PMID 17593171
- [Result] Riddell RH, Goldman H, Ransohoff DF, Appelman HD, Fenoglio CM, Haggitt RC, Ahren C, Correa P, Hamilton SR, Morson BC, et al. Dysplasia in inflammatory bowel disease: standardized classification with provisional clinical applications. Hum Pathol. 1983 Nov;14(11):931-68. doi: 10.1016/s0046-8177(83)80175-0. PMID 6629368
- [Result] Schlemper RJ, Riddell RH, Kato Y, Borchard F, Cooper HS, Dawsey SM, Dixon MF, Fenoglio-Preiser CM, Flejou JF, Geboes K, Hattori T, Hirota T, Itabashi M, Iwafuchi M, Iwashita A, Kim YI, Kirchner T, Klimpfinger M, Koike M, Lauwers GY, Lewin KJ, Oberhuber G, Offner F, Price AB, Rubio CA, Shimizu M, Shimoda T, Sipponen P, Solcia E, Stolte M, Watanabe H, Yamabe H. The Vienna classification of gastrointestinal epithelial neoplasia. Gut. 2000 Aug;47(2):251-5. doi: 10.1136/gut.47.2.251. PMID 10896917
- See also: Related Info — http://www.getaid.org